CLINICAL TRIAL: NCT00611286
Title: PROlonging Dual Antiplatelet Treatment In Patients With Coronary Artery Disease After Graded Stent-induced Intimal Hyperplasia studY
Brief Title: Synergy Between Stent and Drugs to Avoid Ischemic Recurrences After Percutaneous Coronary Intervention
Acronym: PRODIGY
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Marco Valgimigli (Other)
Responsible Party: Sponsor-Investigator, Marco Valgimigli, Head of the Catheterization laboratory, Università degli Studi di Ferrara
Organization: Università degli Studi di Ferrara (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: SSD-03-I
Record Dates: First submitted 2007-12-26; First posted 2008-02-08 (Estimated); Last update posted 2012-10-10 (Estimated); Status verified 2012-10

CONDITIONS: Coronary Artery Disease
Keywords: Drug-eluting stent; clopidogrel; bare metal stent; landmark analysis; Patients with coronary artery disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Purinergic P2Y Receptor Antagonists; Thienopyridines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): treatment with Aspirin and clopidogrel for 24 months after coronary intervention with stents. This group of patients will be randomized in a 1:1:1:1 ratio to receive bare metal stent, Zotarolimus-eluting stent, paclitaxel-eluting stent or everolimus-eluting stent.
  Interventions: Drug: clopidogrel treatment after bare metal stent implantation; Drug: clopidogrel after zotarolimus-eluting stent implantation; Drug: clopidogrel after paclitaxel-eluting stent implantation; Drug: clopidogrel after everolimus-eluting stent implantation
- 2 (Active Comparator): Treatment with aspirin and clopidogrel for minimum 1 or 6 month(s) after BMS or DES implantation, respectively. This group of patients will be randomized in a 1:1:1:1 ratio to receive bare metal stent, Zotarolimus-eluting stent, paclitaxel-eluting stent or everolimus-eluting stent
  Interventions: Drug: clopidogrel treatment after bare metal stent implantation; Drug: clopidogrel after zotarolimus-eluting stent implantation; Drug: clopidogrel after paclitaxel-eluting stent implantation; Drug: clopidogrel after everolimus-eluting stent implantation

INTERVENTIONS:
Drug: clopidogrel treatment after bare metal stent implantation — extending use of clopidogrel on top of aspirin up to 24 months after coronary implantation of bare metal stent
  Other Names: oral ADP receptor blockers; thienopyridines
  Arms: 1
Drug: clopidogrel treatment after bare metal stent implantation — Adding clopidogrel on top of Aspirin according to the practice suggested by Italian national institute of health, i.e. 1 month after BMS implantation.
  Other Names: Oral ADP receptor blocker; thienopyridines
  Arms: 2
Drug: clopidogrel after zotarolimus-eluting stent implantation — extending use of clopidogrel on top of aspirin up to 24 months after coronary implantation of zotarolimus-eluting stent coronary implantation
  Other Names: ADP recepots blockers; p2y12 receptor blockers
  Arms: 1
Drug: clopidogrel after paclitaxel-eluting stent implantation — extending use of clopidogrel on top of aspirin up to 24 months after coronary implantation of paclitaxel-eluting stent
  Other Names: ADP receptor blockers; P2Y12 receptor blocker
  Arms: 1
Drug: clopidogrel after everolimus-eluting stent implantation — extending use of clopidogrel on top of aspirin up to 24 months after coronary implantation of Everolimus-eluting stent
  Other Names: ADP receptor blockers; P2Y12 receptor blocker
  Arms: 1
Drug: clopidogrel after zotarolimus-eluting stent implantation — Adding clopidogrel on top of Aspirin according to the practice suggested by Italian national institute of health, i.e. 6 month after DES implantation.
  Other Names: ADP receptor blockers; P2Y12 receptor blocker
  Arms: 2
Drug: clopidogrel after paclitaxel-eluting stent implantation — Adding clopidogrel on top of Aspirin according to the practice suggested by Italian national institute of health, i.e. 6 month after DES implantation.
  Other Names: ADP receptor blockers; P2Y12 receptor blockers
  Arms: 2
Drug: clopidogrel after everolimus-eluting stent implantation — Adding clopidogrel on top of Aspirin according to the practice suggested by Italian national institute of health, i.e. 6 month after DES implantation.
  Other Names: ADP receptor blockers; P2Y12 receptor blockers
  Arms: 2

SUMMARY:
The duration of dual antiplatelet treatment (i.e. asprin and clopidogrel) after drug-eluting stent implantation is highly debated. This study will evaluate the value of extending such treatment up to 2 years after the procedure as compared to conventional treatment according to our national health institute guidelines (i.e. minimum 1 month after bare metal stent and 6 months after drug-eluting stent) on the composite endpoint of death, MI or stroke.

DETAILED DESCRIPTION:
This is a randomized, multi-center, open-label, study to evaluate the efficacy and safety profile of prolonged dual antiplatelet treatment (i.e. up to 2-year) with aspirin and clopidogrel after coronary stenting compared to currently recommended antiplatelet regimens (i.e. dual antiplatelet treatment for minimum 1 month after BMS or 6 months after DES implantation). As the degree of intimal hyperplasia (IH) suppression provided by the coronary stent system may be expected to influence the comparison between conventional versus prolonged dual antiplatelet treatment (DAT), patients in each group will be further randomized to no (BMS), intermediate (Endeavor), moderately high (Taxus) or very high (Xience V) degree of IH suppression so to minimize the confounding role of IH suppression on the primary hypothesis. Patients will be then follow-up on a clinical basis at 1, 6, 12, 18 and 24 months for the primary hypothesis and then every year up to five for secondary hypotheses.

In the conventional dual antiplatelet therapy group receiving one or more BMS implantation at the time of PCI, length of DAT may be influenced by acuity of clinical presentation. According to the CURE study (JAMA. 2002 Nov 20;288(19):2411-20), patients presenting with non-ST segment elevation acute coronary syndromes may be felt to require longer than 1 month DAT. Thus, to impose 1-month only of DAT duration after PCI may be not regarded as conventional at current stage. Based on this consideration, the protocol will allow extension of DAT up to 6 months after PCI in the conventional BMS group in those patients satisfying the inclusion and exclusion criteria of the CURE study at discretion of the treating physician.Extension of DAt up to 6 months after BMS in patients with STEMI is not recommended byt will be allowed as per protocol

Dual antiplatelet treatment refers to the use of Aspirin at doses ranging from 75 up to 325 mg/day p.o. in conjunction with clopidogrel (75 mg/day). Ticlopidine (250 mg/ twice a day) is a second-choice drug and it will be allowed in cases where clopidogrel is not well tolerated or unavailable. Clopidogrel and ticlopidine are equipotent antiplatelet agents. Both of them belong the class of thienopyridines and they act by inhibiting the the P2Y12 ADP receptor on platelets.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females ≥ 18 years of age with coronary artery disease with low, intermediate or high-risk coronary anatomy, which is considered suitable for PCI with stent placement.
2. Subjects who have provided written informed consent prior to initiation of any study-related procedures, prior to receiving any pre-procedural sedation and who agree to comply with all protocol-specified procedures.

Exclusion Criteria:

1. Women who are pregnant. Women of childbearing potential must have a negative pregnancy test (urine or serum HCG) within 7 days prior to randomization; as close to randomization as possible, within 24 hours preferred.
2. Allergy or intolerance to aspirin, or both clopidogrel and ticlopidine
3. Subjects with a contraindication to anticoagulation and/or increased bleeding risk:

   * Past or present bleeding disorder including a history of the following within 1 month prior to randomization: clinically relevant gastrointestinal bleeding, gross (visible) hematuria,
   * Planned major surgery including CABG after or within 1 month prior to randomization.
   * Any subject with a known coagulopathy, platelet disorder, or history of thrombocytopenia.
4. Subjects with a history of cancer (limiting survival) not known to be disease free, with the exception of basal cell carcinoma of the skin.
5. History of clinically important, recent or ongoing alcohol abuse or other drug abuse.
6. Known platelet count <100,000/mm3 (<100 x 109/L).
7. Subjects who is unable to give informed consent and assurance for complete contact through 2 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1700 (Estimated)
Dates: Start 2006-12; Primary Completion 2010-12 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Composite of death, myocardial infarction or stroke occurring in the time window from 31 days and up to 24 months after intervention. | 24 months

SECONDARY OUTCOMES:
To evaluate the effect of intimal hyperplasia inhibition by drug-release (i.e. different stent types) on the composite of death and myocardial infarction 2 years after intervention | 24 months
Composite of death or myocardial infarction up to 24 months after intervention | 24 months
Cumulative incidence of Stent thrombosis according to the academic consortium definition after 30 days and up to 24 months after intervention | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Marco Valgimigli, MD, PhD, Principal Investigator — University of Ferrara, Italy
Locations (1):
- Azienda Ospedaliera Universitaria di Ferrara, Ferrara, Emilia-Romagna, Italy

REFERENCES:
- [Derived] Natale P, Palmer SC, Saglimbene VM, Ruospo M, Razavian M, Craig JC, Jardine MJ, Webster AC, Strippoli GF. Antiplatelet agents for chronic kidney disease. Cochrane Database Syst Rev. 2022 Feb 28;2(2):CD008834. doi: 10.1002/14651858.CD008834.pub4. PMID 35224730
- [Derived] Gargiulo G, Heg D, Ferrari F, Percoco G, Campo G, Tumscitz C, Colombo F, Zuffi A, Castriota F, Cremonesi A, Windecker S, Valgimigli M. Stent and Dual Antiplatelet Therapy Duration Comparisons in the Setting of a Multicenter Randomized Controlled Trial: Can the Operator Experience Affect the Study Results? J Am Heart Assoc. 2017 Dec 23;6(12):e007150. doi: 10.1161/JAHA.117.007150. PMID 29275371
- [Derived] Piccolo R, Gargiulo G, Franzone A, Santucci A, Ariotti S, Baldo A, Tumscitz C, Moschovitis A, Windecker S, Valgimigli M. Use of the Dual-Antiplatelet Therapy Score to Guide Treatment Duration After Percutaneous Coronary Intervention. Ann Intern Med. 2017 Jul 4;167(1):17-25. doi: 10.7326/M16-2389. Epub 2017 Jun 13. PMID 28605779
- [Derived] Franzone A, Piccolo R, Gargiulo G, Ariotti S, Marino M, Santucci A, Baldo A, Magnani G, Moschovitis A, Windecker S, Valgimigli M. Prolonged vs Short Duration of Dual Antiplatelet Therapy After Percutaneous Coronary Intervention in Patients With or Without Peripheral Arterial Disease: A Subgroup Analysis of the PRODIGY Randomized Clinical Trial. JAMA Cardiol. 2016 Oct 1;1(7):795-803. doi: 10.1001/jamacardio.2016.2811. PMID 27572001
- [Derived] Gargiulo G, Costa F, Ariotti S, Biscaglia S, Campo G, Esposito G, Leonardi S, Vranckx P, Windecker S, Valgimigli M. Impact of proton pump inhibitors on clinical outcomes in patients treated with a 6- or 24-month dual-antiplatelet therapy duration: Insights from the PROlonging Dual-antiplatelet treatment after Grading stent-induced Intimal hyperplasia studY trial. Am Heart J. 2016 Apr;174:95-102. doi: 10.1016/j.ahj.2016.01.015. Epub 2016 Jan 25. PMID 26995375
- [Derived] Costa F, Tijssen JG, Ariotti S, Giatti S, Moscarella E, Guastaroba P, De Palma R, Ando G, Oreto G, Zijlstra F, Valgimigli M. Incremental Value of the CRUSADE, ACUITY, and HAS-BLED Risk Scores for the Prediction of Hemorrhagic Events After Coronary Stent Implantation in Patients Undergoing Long or Short Duration of Dual Antiplatelet Therapy. J Am Heart Assoc. 2015 Dec 7;4(12):e002524. doi: 10.1161/JAHA.115.002524. PMID 26643501
- [Derived] Costa F, Adamo M, Ariotti S, Ferrante G, Navarese EP, Leonardi S, Garcia-Garcia H, Vranckx P, Valgimigli M. Left main or proximal left anterior descending coronary artery disease location identifies high-risk patients deriving potentially greater benefit from prolonged dual antiplatelet therapy duration. EuroIntervention. 2016 Feb;11(11):e1222-30. doi: 10.4244/EIJY15M08_04. PMID 26342472
- [Derived] Costa F, Vranckx P, Leonardi S, Moscarella E, Ando G, Calabro P, Oreto G, Zijlstra F, Valgimigli M. Impact of clinical presentation on ischaemic and bleeding outcomes in patients receiving 6- or 24-month duration of dual-antiplatelet therapy after stent implantation: a pre-specified analysis from the PRODIGY (Prolonging Dual-Antiplatelet Treatment After Grading Stent-Induced Intimal Hyperplasia) trial. Eur Heart J. 2015 May 21;36(20):1242-51. doi: 10.1093/eurheartj/ehv038. Epub 2015 Feb 25. PMID 25718355
- [Derived] Valgimigli M, Tebaldi M, Borghesi M, Vranckx P, Campo G, Tumscitz C, Cangiano E, Minarelli M, Scalone A, Cavazza C, Marchesini J, Parrinello G; PRODIGY Investigators. Two-year outcomes after first- or second-generation drug-eluting or bare-metal stent implantation in all-comer patients undergoing percutaneous coronary intervention: a pre-specified analysis from the PRODIGY study (PROlonging Dual Antiplatelet Treatment After Grading stent-induced Intimal hyperplasia studY). JACC Cardiovasc Interv. 2014 Jan;7(1):20-8. doi: 10.1016/j.jcin.2013.09.008. Epub 2013 Dec 11. PMID 24332420
- [Derived] Campo G, Tebaldi M, Vranckx P, Biscaglia S, Tumscitz C, Ferrari R, Valgimigli M. Short- versus long-term duration of dual antiplatelet therapy in patients treated for in-stent restenosis: a PRODIGY trial substudy (Prolonging Dual Antiplatelet Treatment After Grading Stent-Induced Intimal Hyperplasia). J Am Coll Cardiol. 2014 Feb 18;63(6):506-12. doi: 10.1016/j.jacc.2013.09.043. Epub 2013 Oct 23. PMID 24161321
- [Derived] Valgimigli M, Borghesi M, Tebaldi M, Vranckx P, Parrinello G, Ferrari R; PROlonging Dual antiplatelet treatment after Grading stent-induced Intimal hyperplasia studY Investigators. Should duration of dual antiplatelet therapy depend on the type and/or potency of implanted stent? A pre-specified analysis from the PROlonging Dual antiplatelet treatment after Grading stent-induced Intimal hyperplasia studY (PRODIGY). Eur Heart J. 2013 Mar;34(12):909-19. doi: 10.1093/eurheartj/ehs460. Epub 2013 Jan 12. PMID 23315904
- [Derived] Valgimigli M, Campo G, Monti M, Vranckx P, Percoco G, Tumscitz C, Castriota F, Colombo F, Tebaldi M, Fuca G, Kubbajeh M, Cangiano E, Minarelli M, Scalone A, Cavazza C, Frangione A, Borghesi M, Marchesini J, Parrinello G, Ferrari R; Prolonging Dual Antiplatelet Treatment After Grading Stent-Induced Intimal Hyperplasia Study (PRODIGY) Investigators. Short- versus long-term duration of dual-antiplatelet therapy after coronary stenting: a randomized multicenter trial. Circulation. 2012 Apr 24;125(16):2015-26. doi: 10.1161/CIRCULATIONAHA.111.071589. Epub 2012 Mar 21. PMID 22438530
- [Derived] Valgimigli M, Campo G, Percoco G, Monti M, Ferrari F, Tumscitz C, Zuffi A, Colombo F, Kubbajeh M, Cavazza C, Cangiano E, Tebaldi M, Minarelli M, Arcozzi C, Scalone A, Frangione A, Borghesi M, Marchesini J, Parrinello G, Ferrari R. Randomized comparison of 6- versus 24-month clopidogrel therapy after balancing anti-intimal hyperplasia stent potency in all-comer patients undergoing percutaneous coronary intervention Design and rationale for the PROlonging Dual-antiplatelet treatment after Grading stent-induced Intimal hyperplasia study (PRODIGY). Am Heart J. 2010 Nov;160(5):804-11. doi: 10.1016/j.ahj.2010.07.034. PMID 21095265